CLINICAL TRIAL: NCT03220308
Title: Mindfulness Training for Children With ADHD and Mindful Parenting
Brief Title: Mindfulness Training for Children With Attention-Deficit/Hyperactivity Disorder (ADHD) and Mindful Parenting
Acronym: MindChamp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karakter Kinder- en Jeugdpsychiatrie (Other)
Collaborators: Fonds Psychische Gezondheid (Other); European Commission (Other); UvA minds (Unknown); Radboud University Medical Center (Other); University of Amsterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20016 MIND
Record Dates: First submitted 2017-06-20; First posted 2017-07-18 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Self-control; Well-being
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Self-Control | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care-as-usual (CAU) only (Other): Care-as-usual for children (8-16 years old) with ADHD
  Interventions: Other: Care-as-usual for children (8-16 years old) with ADHD
- Mindfulness for child and parent + CAU (Experimental): MYmind mindfulness training in addition to care-as-usual for children aged 8-16 years with ADHD
  Interventions: Other: MYmind mindfulness training; Other: Care-as-usual for children (8-16 years old) with ADHD

INTERVENTIONS:
Other: MYmind mindfulness training — The MYmind mindfulness training uses a standardised protocol based on mindfulness-based cognitive therapy. It consists of 8 weekly group sessions of 90 minutes for youth with ADHD, and parallel mindful parenting training for the parents. Eight weeks after the last session there is a single 90 minutes booster session.
  Other Names: Mindfulness for children with ADHD and mindful parenting
  Arms: Mindfulness for child and parent + CAU
Other: Care-as-usual for children (8-16 years old) with ADHD — According to the Dutch Multidisciplinary guidelines for the diagnosis and treatment of ADHD, care-as-usual for children aged 8-16 years with ADHD consists of psycho-education and the prescription of medication approved for ADHD and/or evidence-based parent and/or teacher-administered behaviour therapy, preferably both medication and behaviour therapy. First-line option for medication is a psychostimulant, second-line option is atomoxetine, and third-line options are alpha-2 presynaptic agonists or tricyclic antidepressants (imipramine).

SUMMARY:
This study evaluates the effectiveness of an 8-week mindfulness group training for children (8-16 years old) with ADHD in combination with a parallel mindful parenting training for their parents. Half of the participants will be randomly assigned to the mindfulness training in addition to care-as-usual (CAU); the other half to CAU-only.

The hypothesis is that compared to care-as-usual only, the addition of the mindfulness training will improve self-control of youth with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Child has a clinical diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Disorders; DSM-IV or DSM-5 system, and confirmed by a structured interview (The Schedule for Affective Disorders and Schizophrenia for school-Age Children (K-SADS)).
* Child receives CAU and has remaining ADHD-symptoms (average score > 1.0 on the investigator-rated DSM-5 items from the Conners' ADHD rating scale).
* Child is between 8 and 16 years old.
* At least one parent is willing to participate.
* ADHD medication dose is stable, or there is an informed decision on not taking ADHD medication.
* Psychiatric comorbidities are allowed except psychosis, bipolar illness, active suicidality, untreated posttraumatic stress disorder or substance use, provided ADHD is the primary diagnosis in the child; similarly, psychopathology in the parents is allowed except psychosis, bipolar disorder, active suicidality, untreated posttraumatic stress disorder or substance use.
* Child and parent have an estimated intelligence quotient (IQ) ≥ 80.
* Child and parent have adequate mastery of Dutch language.

Exclusion Criteria:

* Child or the participating parent(s) have participated in a mindfulness programme in the past year or ever in a Mindful Parenting training.
* Child or parent is participating in another intervention study.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in parent-rated self-control of the child | Baseline, 3, 5 and 9 months
  Behaviour Rating Inventory of Executive Function, parent-report (BRIEF-P)

SECONDARY OUTCOMES:
Change from Baseline in parent-rated behaviour problems of the child | Baseline, 3, 5 and 9 months
  Conners' Parent Rating Scales-Revised: Long (CPRS-R), subscales: inattentive and hyperactive-impulsive symptoms according to the 4th version of the Diagnostic and Statistical Manual (DSM-IV), oppositional, anxious/shy, social problems and the Emotional Lability index
Change from Baseline in parent-rated autistic social impairment of the child | Baseline, 3 and 9 months
  Social Responsiveness Scale, parent-report (SRS-P)
Change from Baseline in parent-rated quality of life of the child | Baseline, 3 and 9 months
  KIDSCREEN-10, parent-report
Change from Baseline in teacher-rated self-control of the child | Baseline, 3 and 5 months
  Behaviour Rating Inventory of Executive Function, teacher-report (BRIEF-T)
Change from Baseline in teacher-rated behaviour problems of the child | Baseline, 3 and 5 months
  Conners' Teacher Rating Scales-Revised: Long (CTRS-R), subscales: inattentive and hyperactive-impulsive symptoms according to the 4th version of the Diagnostic and Statistical Manual (DSM-IV), oppositional, anxious/shy, social problems and the Emotional Lability index
Change from Baseline in teacher-rated autistic social impairment of the child | Baseline and 3 months
  Social Responsiveness Scale, teacher-report (SRS-T)
Change from Baseline in self-rated dispositional mindfulness of the child | Baseline, 3, 5 and 9 months
  Child and Adolescent Mindfulness Measure (CAMM), self-report
Change from Baseline in self-rated brooding of the child | Baseline, 3 and 9 months
  Ruminative Response Scale (RRS), subscale: brooding, self-report
Change from Baseline on the Stop task in the child | Baseline, 3 and 9 months
  Computer based neurocognitive assessments of self-control in the child
Change from Baseline on the Probabilistic reversal learning task in the child | Baseline, 3 and 9 months
  Computer based neurocognitive assessments of self-control in the child
Change from Baseline on the Temporal discounting task in the child | Baseline, 3 and 9 months
  Computer based neurocognitive assessments of self-control in the child
Change from Baseline in self-rated self-control of the parent | Baseline, 3, 5 and 9 months
  Behaviour Rating Inventory of Executive Function, self-report (BRIEF-A)
Change from Baseline in self-rated ADHD traits of the parent | Baseline, 3, 5 and 9 months
  DSM-5 based ADHD traits, self-report
Change from Baseline in self-rated mindfulness in parenting of the parent | Baseline, 3, 5 and 9 months
  Interpersonal Mindfulness in Parenting Scale (IM-P), self-report
Change from Baseline in self-rated autistic traits of the parent | Baseline, 3 and 9 months
  Short Autism Quotient Questionnaire-Adult Version (AQ-10), self-report
Change from Baseline in self-rated symptoms of depression, anxiety and stress in the parent | Baseline, 3 and 9 months
  Depression Anxiety Stress Scale-21 (DASS-21), self-report
Change from Baseline in self-rated emotional well-being, psychological well-being and social well-being of the parent | Baseline, 3 and 9 months
  Mental Health Continuum-Short Form (MHC-SF), self-report
Change from Baseline in self-rated quality of life of the parent | Baseline, 3 and 9 months
  World Health Organization-Five Well-Being Index (WHO-5), self-report
Change from Baseline in self-rated brooding of the parent | Baseline, 3 and 9 months
  Ruminative Response Scale (RRS), subscale: brooding, self-report
Change from Baseline on the Stop task in the parent | Baseline, 3 and 9 months
  Computer based neurocognitive assessments of self-control in the parent
Change from Baseline on the Probabilistic reversal learning task in the parent | Baseline, 3 and 9 months
  Computer based neurocognitive assessments of self-control in the parent
Change from Baseline on the Temporal discounting task in the parent | Baseline, 3 and 9 months
  Computer based neurocognitive assessments of self-control in the parent

CONTACTS AND LOCATIONS:
Overall Officials: Jan K Buitelaar, Principal Investigator — Karakter Kinder- en Jeugdpsychiatrie
Locations (3):
- Netherlands (3):
  - Karakter, Expertisecentrum voor kinder- en jeugdpsychiatrie, Arnhem, Gelderland
  - Karakter, Expertisecentrum voor kinder- en jeugdpsychiatrie, Ede, Gelderland
  - Karakter, Expertisecentrum voor kinder- en jeugdpsychiatrie, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: Yes
Data will be available 18 months after finishing the study. The investigators will give limited access to the data, that is, data can be obtained provided that the applicant will submit a research plan and the investigator of the current study will be involved in the research on the shared data. Data will be anonymised and accompanied by the present study protocol and data list description. Other researchers can contact Karakter (sponsor of the study) to obtain data:
  Address: Reinier Postlaan 12 6525 GC Nijmegen Phone: 024 351 22 22 Email: info.nijmegen@karakter.com

REFERENCES:
- [Background] Siebelink NM, Bogels SM, Boerboom LM, de Waal N, Buitelaar JK, Speckens AE, Greven CU. Mindfulness for children with ADHD and Mindful Parenting (MindChamp): Protocol of a randomised controlled trial comparing a family Mindfulness-Based Intervention as an add-on to care-as-usual with care-as-usual only. BMC Psychiatry. 2018 Jul 25;18(1):237. doi: 10.1186/s12888-018-1811-y. PMID 30045714
- See also: recruitment text (Dutch) — http://www.google.nl/url?sa=t&rct=j&q=&esrc=s&source=web&cd=25&cad=rja&uact=8&ved=0ahUKEwjJzP3slp_UAhXRZFAKHQ0zB3s4FBAWCEgwBA&url=http%3A%2F%2Fwww.ru.nl%2Fpublish%2Fpages%2F829896%2Fmindchamp.pdf&usg=AFQjCNErU__IASzNyGwRKHOeb2c-Qk5r8g
- See also: recruitment text (Dutch) — http://www.adhdnetwerk.nl/ADHD.aspx?id=481&idn=450
- See also: abstract for symposium (English) — https://www.radboudcentrumvoormindfulness.nl/wp-content/uploads/2016/02/Mindfulness-with-children-with-ADHD-potential-working-mechanisms-Corina-Greven-Nienke-Siebelink.pdf
- See also: blog post on the feasibility of the study (English) — https://mind-the-gap.live/2017/01/31/mindfulness-for-children-with-adhd-is-that-possible/